CLINICAL TRIAL: NCT01229280
Title: Comparative Bioavailability of Darifenacin Extended Release Oral Formulation [Darisec(R)7.5 mg vs. Enablex(R)7.5 mg]: Single-dose, Postprandial State, Randomized, Two-sequence, Two-period, Crossover Study in Healthy Volunteers.
Brief Title: Single Dose Bioequivalence Study of Darifenacin Tablets 7.5 mg in Fed Healthy Volunteers.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Center for Clinical Pharmacology Research Bdbeq S.A. (Other)
Collaborators: Laboratorio Elea Phoenix S.A. (Industry)
Responsible Party: Francisco E. Estevez-Carrizo, Center for Clinical Pharmacology Research Bdbeq S.A.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BDBEQ_DFNLP/ELEA_010
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2010-10

CONDITIONS: Bioequivalency
Keywords: Bioequivalence; Darifenacin; Healthy volunteers; Postprandial
MeSH Terms: interventions — darifenacin; Muscarinic Antagonists; Cholinergic Antagonists; Cholinergic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Darisec(R) 7.5 mg (Experimental)
  Interventions: Drug: Darifenacin
- Enablex(R) 7.5 mg (Active Comparator)
  Interventions: Drug: Darifenacin

INTERVENTIONS:
Drug: Darifenacin — Single dose 7.5 mg tablets of darifenacin
  Other Names: Muscarinic antagonist; Cholinergic antagonist; Cholinergic agent; Darisec
  Arms: Darisec(R) 7.5 mg
Drug: Darifenacin — Single dose 7.5 mg tablets of Darifenacin
  Other Names: Muscarinec antagonist; Cholinergic antagonist; Cholinergic agent; Enablex
  Arms: Enablex(R) 7.5 mg

SUMMARY:
The proposed study was designed as a randomized two-sequence, two period crossover trial to assess the bioequivalence, pharmacokinetic profiling and safety of a brand generic formulation of darifenacin [Darisec(R) 7.5 mg] vs. the innovator [Enablex(R)7.5 mg]in healthy volunteers in postprandial state.

DETAILED DESCRIPTION:
Darifenacin is a muscarinic receptor antagonist drug used to treat overactive bladder. There is a new formulation of darifenacin extended release developed by an argentinian pharmaceutical company. A bioequivalence study will be performed to validate pharmaceutical development before introducing the product in the market.

The purpose in this study is to evaluate the relative bioavailability, pharmacokinetic profiling and safety of a brand generic formulation of darifenacin [Darisec(R) 7.5 mg] vs. the innovator [Enablex(R) 7.5 mg]in 24 healthy uruguayan volunteers after a high fat breakfast of 1000 calories (50% fat, 35% carbohydrates, and 15% proteins)to establish their average bioequivalence.

The bioequivalence will be evaluated using:

* The Area Under the Curve (AUC),
* The peak plasma concentration (Cmax).

The pharmacokinetic characteristics of the drug formulations will be described calculating:

* The time to peak concentration (Tmax)
* The elimination constant (Ke)
* The elimination half-life (t1/2e)
* The systemic clearance (Cls)

Safety will be evaluated recording:

* Reported adverse events
* Vital signs (blood pressure, heart rate, body temperature)
* Laboratory analysis (hemogram, hepatic enzymes, creatinine, sugar in blood, etc.)
* EKG and chest XRays

Bioequivalence will be claimed if the drugs comply with local and FDA regulatory requirements:

* Mean AUCt/AUCr and 90% confidence interval within 0.80-1.25
* Mean Cmaxt/Cmaxr and 90% confidence interval within 0.80-1.25

Pharmacokinetic profiling will be evaluated by describing the pharmacokinetic characteristics of both drug in adequate two-way tables.

Safety will be evaluated comparing incidence of adverse events/adverse effects for both products.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects 18 to 50 years of age (inclusive).
* In good health, as determined by lack of clinically significant abnormalities at screening as judged by the physician.
* Female subjects are required to use a medically accepted method of hormonal contraception or abstinence throughout the entire study period and for one week after the study is completed.
* Body mass index within the range of 18.5 and 29.9 kg/m2 and weight at least 45 kg.

Exclusion Criteria:

* Known hypersensitivity or severe adverse event to darifenacin or similar drugs.
* Urinary, retention, narrow-angle glaucoma, myasthenia gravis, severe hepatic impairment, severe ulcerative colitis, toxic megacolon.
* Symptomatic hiatus hernia, erosive or symptomatic gastroesophageal reflux disease/heartburn (>2 days in a week), severe constipation, gastrointestinal obstructive disorder, and gastric retention.
* Clinically significant cardiac abnormalities, fainting, low blood pressure upon standing, irregular heartbeats.
* Acute or chronic bronchospastic disease(including asthma and Chronic Obstructive Pulmonary Disease).
* Clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis).
* Smokers of more than 5 cigarettes a week.
* Regular use of any drug known to induce or inhibit hepatic drug metabolism (particularly those that affect CYP2D6) within 30 days prior to each study drug administration.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs which may jeopardize participation in the study.
* Immunodeficiency diseases, including a positive HIV (Elisa or Western blot) test result.
* Positive Hepatitis B Surface antigen (HBsAg) or Hepatitis C results.
* Drug or alcohol abuse within the 6 months prior to dosing.
* Use of prescription drugs within 1 month prior to dosing, or over-the-counter medication (vitamins, herbal supplements, dietary supplements)within 2 weeks prior to dosing. Paracetamol and ibuprofen are acceptable.
* Participation in any clinical investigation within 12 weeks prior to dosing.
* Donation or loss of 400 ml or more of blood within 8 weeks prior to dosing.
* Significant illness within 2 weeks prior to dosing.
* Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-01 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Extent of absorption | 72 hours
  Extent of absorption will be measured using the area under the plasma concentration of darifenacin vs time from time 0 to the last sample point (AUC0-t) and from time 0 to infinity (AUC0-inf.
Rate of absorption | 72
  Rate of abosorption will be measured using peak concentration of darifenacin (Cmax)taken from the concentration vs. time curve.

SECONDARY OUTCOMES:
Time to peak concentration (tmax) | 72
  Tmax is the time elapsed from ingestion of darifenacin tablets to plasma peak concentration (Cmax)
Elimination rate constant (Ke) | 72 hours
  The elimination rate constant is the fractional rate of drug disappearance form the peripheral compartement, measured in the log-linear elimination phase.
Elimination Half-life (t1/2e) | 72 hours
  t1/2e is the time in which the concentration in the log-linear elimination phase drops by half.
Systemic clearance (Cls) | 72 hours
  Cls is the amount of plasma volume units that are totally cleared of the drug in the unit of time.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco E. Estevez-Carrizo, MD, Study Director — Univerisity of Montevideo. Biomedical Science Center.Prudencio de Pena 2440, 11600 Montevideo. Uruguay; Susana Parrillo, M.D., Principal Investigator — Center for Clinical Pharmacology Research Bdbeq S.A., Br. Artigas 1632. c.p. 11600 Montevideo. Uruguay.
Locations (1):
- Center for Clinical Pharmacology Research (CCPR) Bdbeq S.A. Hospital Italiano., Montevideo, Montevideo Department, Uruguay

REFERENCES:
- [Background] Skerjanec A. The clinical pharmacokinetics of darifenacin. Clin Pharmacokinet. 2006;45(4):325-50. doi: 10.2165/00003088-200645040-00001. PMID 16584282
- [Background] Croom KF, Keating GM. Darifenacin: in the treatment of overactive bladder. Drugs Aging. 2004;21(13):885-92; discussion 893-4. doi: 10.2165/00002512-200421130-00005. PMID 15493952
- [Background] Staskin DR. Overactive bladder in the elderly: a guide to pharmacological management. Drugs Aging. 2005;22(12):1013-28. doi: 10.2165/00002512-200522120-00003. PMID 16363885
- [Background] Kerbusch T, Wahlby U, Milligan PA, Karlsson MO. Population pharmacokinetic modelling of darifenacin and its hydroxylated metabolite using pooled data, incorporating saturable first-pass metabolism, CYP2D6 genotype and formulation-dependent bioavailability. Br J Clin Pharmacol. 2003 Dec;56(6):639-52. doi: 10.1046/j.1365-2125.2003.01967.x. PMID 14616424
- [Background] Dmochowski RR, Appell RA. Advancements in pharmacologic management of the overactive bladder. Urology. 2000 Dec 4;56(6 Suppl 1):41-9. doi: 10.1016/s0090-4295(00)01020-7. PMID 11114562